CLINICAL TRIAL: NCT02225431
Title: Personalized Versus Standard Hydration for Prevention of Contrast Induced Acute Kidney Injury. A Randomized Trial With Bioimpedance Analysis.
Brief Title: Personalized Versus Standard Hydration for Prevention of CI-AKI: a Randomized Trial With Bioimpedance Analysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale Misericordia e Dolce (Other)
Responsible Party: Principal Investigator, Mauro Maioli, MD, Ospedale Misericordia e Dolce
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Prato0706; 2013/1
Record Dates: First submitted 2014-08-24; First posted 2014-08-26 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Acute Kidney Injury
Keywords: Contrast-induced nephropathy; Contrast-Induced acute kidney injury; Contrast media; Angiography; Coronary percutaneous intervention
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard saline infusion (Active Comparator): All patients received standard intravenous saline hydration (0.9% sodium chloride, 1 ml/kg/h for 12 hours before and after procedure)
  Interventions: Drug: sodium chloride infusion
- Double saline infusion (Experimental): All patients received double dose of intravenous saline hydration (0.9% sodium chloride, 2 ml/kg/h for 12 hours before and after procedure)
  Interventions: Drug: sodium chloride infusion

INTERVENTIONS:
Drug: sodium chloride infusion

SUMMARY:
The aim of this study was to evaluate, in patients with "lower fluid status" defined by bioimpedance analysis, whether two different protocol of IV isotonic saline infusion are associated with different volume expansion and differing risks for CI-AKI in patients undergoing coronary angiographic procedures.

DETAILED DESCRIPTION:
Iodinated contrast media are a well-recognized cause of iatrogenic acute kidney injury in patients undergoing imaging diagnostic or therapeutic procedures (contrast-induced acute kidney injury, CI-AKI).

Several protocols have been tested for the prevention of CI-AKI, including periprocedural hydration with isotonic saline or sodium bicarbonate, antioxidant compounds, use of low- or iso-osmolar contrast agents, and hemofiltration or dialysis. The results of these interventions and strategies have been often disappointing or inconclusive and intravenous volume expansion remains the only therapy of undisputed efficacy.

Bioimpedance analysis is an inexpensive, rapid, and accurate tool for evaluating a patient's hydration status, and can be performed at the bedside within minutes [Maioli, JACC 1014;63:1387-94]. In this study we defined patients with "lower fluid status" with high risk of CI-AKI (Male with resistance/height ratio > 315 Ohm/meter and Female > 380 Ohm/meter). BIVA may represent the optimal tool to monitor the adequacy of volume expansion and protective strategy delivery.

However, most hydration protocols rely on a "one size fits all" approach with a fixed volume and time of infusion without an assessment of whether adequate hydration was achieved. This practice risks either under-hydration without true amelioration of CI-AKI risk or over-hydration with risk of adverse outcomes.

Thus, on the basis of results of BIVA testing a randomized fluid infusion plan is prescribed.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients admitted in Cardiology Unit for coronary or peripheral angiography with "lower fluid status" defined on the basis bio-impedance analysis (Male with resistance/height ratio > 315 Ohm/meter and Female > 380 Ohm/meter).

Exclusion Criteria:

* contrast medium administration within the 10 days
* end stage renal failure requiring dialysis
* refused to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2012-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Incidence of contrast-induced acute kidney injury | 1 day
  contrast acute kidney injury is defined as an increase in serum Cystatin C concentration 10% above the baseline value at 24 hours after administration of contrast medium

SECONDARY OUTCOMES:
Adverse clinical events | 1 month
  adverse clinical events within 1 month including in-hospital death and need for dialysis or hemofiltration

OTHER OUTCOMES:
Incidence of contrast-induced acute kidney injury | 2 days
  Contrast-induced acute kidney injury defined as an increase in serum creatinine >= 0.3 mg/dl over baseline value within 2 days after the administration of contrast medium

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Maioli, MD, Principal Investigator — Ospedale S. Stefano - Prato - Italy
Locations (1):
- Ospedale Santo Stefano, Prato, Prato, Italy

REFERENCES:
- [Background] Maioli M, Toso A, Leoncini M, Musilli N, Bellandi F, Rosner MH, McCullough PA, Ronco C. Pre-procedural bioimpedance vectorial analysis of fluid status and prediction of contrast-induced acute kidney injury. J Am Coll Cardiol. 2014 Apr 15;63(14):1387-94. doi: 10.1016/j.jacc.2014.01.025. Epub 2014 Feb 12. PMID 24530668
- [Derived] Maioli M, Toso A, Leoncini M, Musilli N, Grippo G, Ronco C, McCullough PA, Bellandi F. Bioimpedance-Guided Hydration for the Prevention of Contrast-Induced Kidney Injury: The HYDRA Study. J Am Coll Cardiol. 2018 Jun 26;71(25):2880-2889. doi: 10.1016/j.jacc.2018.04.022. PMID 29929610